CLINICAL TRIAL: NCT06881433
Title: Immune Checkpoint Inhibitors and Anti-vascular Endothelial Growth Factor Antibody/tyrosine Kinase Inhibitors with or Without Hepatic Arterial Infusion Chemotherapy As First-line Treatment for Advanced Hepatocellular Carcinoma
Brief Title: Immune Checkpoint Inhibitors and Anti-vascular Endothelial Growth Factor Antibody/tyrosine Kinase Inhibitors with or Without HAIC for Advanced HCC
Status: Recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Other Study IDs: CHANCE2504
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: hepatocellular carcinoma; immune checkpoint inhibitors; molecular target therapies; hepatic infusion chemotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Tyrosine kinase inhibitors (TKIs) plus programmed death-1 (PD-1) inhibitors are recommended for patients with advanced hepatocellular carcinoma (HCC) in China. However, these treatments have limited survival benefit in patients with advanced HCC. We aimed to investigate whether hepatic arterial infusion chemotherapy (HAIC) in combination with TKIs and PD-1 inhibitors could improve the efficacy.

DETAILED DESCRIPTION:
The multiple real-world studies have shown that Tyrosine kinase inhibitors (TKIs) plus programmed death-1 (PD-1) inhibitors (TKIs-P) does not result in a high response rate or extended survival for patients with extrahepatic metastases, with an objective response rate (ORR) of less than 20%. Therefore, there is an urgent need to explore effective therapeutic strategies that can enhance the combined antitumor efficacy of TKIs-P and improve the prognosis of patients with advanced hepatocellular carcinoma (HCC). In addition to TKIs-P, more aggressive treatments, such as hepatic arterial infusion chemotherapy (HAIC), have been adopted in the Asia-Pacific region. HAIC significantly increases drug concentration in HCC tissues while decreasing drug distribution in the peripheral blood, thereby improving intrahepatic tumor control and reducing systemic adverse events (AEs). Recent significant advancements have been reported in both local-regional and systemic therapies. Furthermore, the combination of HAIC with TKIs-P (HAIC-TKIs-P) may provide potential synergistic anticancer activity for HCC based on the following rationale: HAIC can effectively kill tumors while promoting the release of tumor antigens, thus transforming "cold tumors" into "hot tumors." At the same time, TKIs can reverse the tumor neovascularization induced by interventional therapies and enhance tumor vasculature normalization. However, it remains unclear whether patients with advanced HCC can benefit from HAIC-TKIs -P through intrahepatic lesion control, thereby impeding tumor progression. Accordingly, this national multiple-centers retrospective study aims to compare the clinical benefits and tolerability of HAIC-TKIs-P versus TKIs-P alone.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of HCC confirmed by radiology, histology, or cytology;
2. Barcelona Clinic Liver Cancer (BCLC) stage B/C;
3. Has not received any previous systemic therapy for HCC (including chemotherapy, molecularly targeted therapy, immunotherapy);
4. Both PD-1/PD-L1 inhibitors and anti-angiogenesis drugs patients received only include marketed drugs but are not limited to HCC approval;
5. HAIC was performed after the first PD-1/PD-L1 inhibitor/anti-angiogenic drug treatment or before treatment (within 3 months);
6. Received at least 1 cycle of PD-1/PD-L1 inhibitor/anti-angiogenic drug combination therapy after HAIC treatment;
7. Has repeated measurable intrahepatic lesions;

Exclusion Criteria:

1. Cholangiocarcinoma, fibrolamellar, sarcomatoid hepatocellular carcinoma, and mixed hepatocellular/cholangiocarcinoma subtypes(confirmed by histology, or pathology) are not eligible;
2. Unable to meet criteria of combination timeframe described above;
3. Child-Pugh C or PS>2 or Severe hepatic encephalopathy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable HCC who received HAIC in combination with PD-1/PD-L1 inhibitors and molecular target therapies under real-world practice conditions
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | up to approximately 2 years
  The OS is defined as the time from the initiation of any combination treatment to death due to any cause.
Progression free survival(PFS) per RECIST 1.1 or mRECIST | up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to RECIST 1.1 or mRECIST) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective response rate(ORR) per RESCIST 1.1 | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per RECIST 1.1.
ORR per mRECIST | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented CR or PR per mRECIST.
Adverse event(AE) per Common Terminology Criteria for Adverse Events(CTCAE) 5.0 | up to approximately 2 years
  The percentage and degree of patients who experience at least one AE, whether or not considered related to the treatment, according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-jun Teng, M.D, Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China